CLINICAL TRIAL: NCT02412150
Title: Effect of Dexmedetomidine Infusion for Postoperative Outcome and Smooth Emergence After Thyroidectomy
Brief Title: Effect of Dexmedetomidine After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Jung, Assist Professor, Chosun University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEX_ENT; 2014-04-004-003 (Other: ChounUHIRB)
Record Dates: First submitted 2015-03-31; First posted 2015-04-09 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Thyroid Tumor
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Desflurane; Gas Scavengers; Remifentanil; Analgesics, Opioid; Thyroidectomy; Surgical Procedures, Operative; Hemodynamics; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Group D) (Experimental): After induction of anesthesia, anesthesia is maintained with desflurane and remifentanil during thyroidectomy.
  Fifteen minutes before the end of surgery, infusion of remifentanil for surgery is discontinued.
  Then, dexmedetomidine has started infusion for 15 min (rate of 0.6 ug/kg/hr). Vital signs and complications of testing drugs are measured before and after infusion of testing drugs.
  Five minutes before the end of surgery, anesthetic gas (desflurane) is discontinued.
  After patient has awake, extubation has done. Extubation time and Recovery time,Cough reflex,Ramsay Sedation Scale, Visual analogue scale, and surgical outcomes such as postoperative bleeding, time to remove drainage and duration of hospital staying, postoperative complications are measured until POD#3.
  Interventions: Drug: Desflurane; Drug: Remifentanil; Procedure: Thyroidectomy; Other: Vital signs; Behavioral: Cough reflex; Behavioral: Ramsay Sedation Scale; Other: Extubation time and Recovery time; Behavioral: Visual analogue scale; Other: Postoperative bleeding; Other: Postoperative complications; Other: Time to remove drainage and duration of hospital staying; Drug: Dexmedetomidine
- Normal Saline (Group N) (Placebo Comparator): After induction of anesthesia, anesthesia is maintained with desflurane and remifentanil during thyroidectomy.
  Fifteen minutes before the end of surgery, infusion of remifentanil for surgery is discontinued. Then, normal saline has started infusion for 15 min (same rate as Group D). Vital signs and complications of testing drugs are measured before and after infusion of testing drugs.
  Five minutes before the end of surgery, anesthetic gas (desflurane) is discontinued.
  After patient has awake, extubation has done. Extubation time and Recovery time,Cough reflex,Ramsay Sedation Scale, Visual analogue scale, and surgical outcomes such as postoperative bleeding, time to remove drainage duration of hospital staying, postoperative complications are measured until POD#3.
  Interventions: Drug: Desflurane; Drug: Remifentanil; Procedure: Thyroidectomy; Other: Vital signs; Behavioral: Cough reflex; Behavioral: Ramsay Sedation Scale; Other: Extubation time and Recovery time; Behavioral: Visual analogue scale; Other: Postoperative bleeding; Other: Postoperative complications; Other: Time to remove drainage and duration of hospital staying; Drug: Normal saline

INTERVENTIONS:
Drug: Desflurane — Anesthesia is maintained with desflurane
  Other Names: Anesthetic gas
Drug: Remifentanil — Remifentanil is infused for the maintenance of anesthesia during surgery and discontinued 15 min before end of surgery
  Other Names: Opioid
Procedure: Thyroidectomy — The aim of this study is evaluation of effect of dexmedetomidine on emergence response and postoperative outcome after thyroidectomy
  Other Names: Surgery
Other: Vital signs — Systolic blood pressure, diastolic blood pressure, mean arterial pressure, and heart rate are measured before infusion of testing drugs, after infusion of them (5 min, 10 min, and 15 min), during extubation (0 min and 5 min after extubation), and at recovery room.
  And the complications such as hypotension, hypertension, bradycardia, tachycardia, and desaturation after infusion of testing drugs are observed.
  Other Names: Hemodynamics
Behavioral: Cough reflex — During recovery from anesthesia at operation room, cough reflex is measured and rated. [Grade 0, no cough; Grade 1, single cough with mild severity; Grade 2, cough persistence less than 5 s with moderate severity; Grade 3, severe, persistent cough for more than 5 s (bucking)]
Behavioral: Ramsay Sedation Scale — When the patient has fully awaken and transferred to the recovery room, Ramsay Sedation Scale is measured.
  1. Awake Patient anxious and agitated or restless or both!
  2. Patient cooperative, oriented and tranquil!
  3. Patient responds to commands only!
  4. Asleep A brisk response to a light glabellar tap or loud auditory stimulus!
  5. A sluggish response to a light glabellar tap or loud auditory stimulus!
  6. No response to a light glabellar tap or loud auditory stimulus
  Other Names: RSS
Other: Extubation time and Recovery time — The time from discontinuing anesthetic gas to endotracheal extubation is measured.
  And the time from the discontinuing of anesthetic gas to transferring to the recovery room is also measured.
Behavioral: Visual analogue scale — The severity of pain after surgery is measured by VAS (at recovery room, POD 1, POD 2, and POD 3)
  Other Names: VAS
Other: Postoperative bleeding — The amount of postoperative bleeding which is collected in the barovac is measured.
Other: Postoperative complications — Postoperative complications after thyroidectomy such as hoarseness and hematoma, and reoperation due to such complication is observed.
Other: Time to remove drainage and duration of hospital staying — The time from the end of surgery to remove drainage is measured. And the duration of hospital staying is measured.
Drug: Dexmedetomidine — Dexmedetomidine has started infusion for 15 min (rate of 0.6 ug/kg/hr) before end of surgery as experimental intervention
  Other Names: Precedex
  Arms: Dexmedetomidine (Group D)
Drug: Normal saline — Normal saline has started infusion for 15 min (as same rate of dexmedetomidine) before end of surgery as control intervention
  Other Names: NS
  Arms: Normal Saline (Group N)

SUMMARY:
The purpose of the present study was to compare the effect of dexmedetomidine which is administered during emergence in adult patients undergoing elective thyroidectomy on smooth emergence form general anesthesia (reducing agitation or coughing, signs of hypertension or tachycardia, or etc.) and postoperative outcome (postoperative bleeding and hospital staying).

DETAILED DESCRIPTION:
Smooth emergence from general anaesthesia after surgery is important to prevent potentially dangerous effects such as hypertension, tachycardia, myocardial ischaemia, arrhythmias and increased intracranial and intra-abdominal pressure. After thyroidectomy, activities during emergence such as agitation or coughing, signs of hypertension or tachycardia, or etc. may lead to postoperative bleeding, resulting in acute airway obstruction or reoperation.

The purpose of the present study was to compare the effect of dexmedetomidine which is administered during emergence in adult patients undergoing elective thyroidectomy on smooth emergence form general anesthesia and postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Female patient,
* Aged 20-60 yr,
* ASA physical status 1-2,
* Patients undergoing elective thyroidectomy under general anesthesia

Exclusion Criteria:

* Sighs of difficult airway,
* History of respiratory disease or chronic cough,
* Cardiovascular disease,
* Pregnant or breast-feeding woman

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2014-04; Primary Completion 2020-11-21 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding | From the end of surgery to the 3rd postoperative day (an expected average of 3 days)
  Postoperative bleeding: Sum of bleeding via barovac

SECONDARY OUTCOMES:
Ramsay Sedation scale | During the recovery time of anesthesia, an expected average of 20 min
  Ramsay Sedation scale at recovery room
Extubation time | During the recovery time of anesthesia, an expected average of 20 min
  time to extubation from the end of surgery
Recovery time of anesthesia | During the recovery time of anesthesia, an expected average of 20 min
  time to transfer to recovery room from the end of surgery
Duration of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Duration of hospital stay
Pain score | From the end of surgery to the 3rd postoperative day (an expected average of 3 days)
  Pain score: NRS
Incidence of postoperative complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Hoarseness, hematoma, and reoperation
Coughing Response | During the recovery time of anesthesia, an expected average of 20 min
  Coughing Response during recovery from anesthesia

OTHER OUTCOMES:
Vital signs | From 15 min before the end of surgery to the time when the patient has transferred to the recovery room, an expected average of 40 min
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure, and heart rate
Complications of testing drug | During infusion of testing drug (15 min)
  Hypertension, hypotension, bradycardia, tachycardia, and desaturation after infusion of dexmedetomidine or normal saline

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Jung, M.D., Study Chair — Chosun University Hospital
Locations (1):
- Chosun University Hospital, Gwangju, Donggu, South Korea

REFERENCES:
- [Background] Patel A, Davidson M, Tran MC, Quraishi H, Schoenberg C, Sant M, Lin A, Sun X. Dexmedetomidine infusion for analgesia and prevention of emergence agitation in children with obstructive sleep apnea syndrome undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Oct;111(4):1004-10. doi: 10.1213/ANE.0b013e3181ee82fa. Epub 2010 Aug 12. PMID 20705788
- [Background] Reeve T, Thompson NW. Complications of thyroid surgery: how to avoid them, how to manage them, and observations on their possible effect on the whole patient. World J Surg. 2000 Aug;24(8):971-5. doi: 10.1007/s002680010160. PMID 10865043
- [Result] Lee B, Lee JR, Na S. Targeting smooth emergence: the effect site concentration of remifentanil for preventing cough during emergence during propofol-remifentanil anaesthesia for thyroid surgery. Br J Anaesth. 2009 Jun;102(6):775-8. doi: 10.1093/bja/aep090. Epub 2009 May 2. PMID 19411668
- [Derived] Kim SH, Kim YS, Kim S, Jung KT. Dexmedetomidine decreased the post-thyroidectomy bleeding by reducing cough and emergence agitation - a randomized, double-blind, controlled study. BMC Anesthesiol. 2021 Apr 12;21(1):113. doi: 10.1186/s12871-021-01325-6. PMID 33845761